CLINICAL TRIAL: NCT05784246
Title: A Multicenter, Phase 3, Open-Label Study to Investigate the Efficacy, Pharmacokinetics, and Safety of Mirikizumab in Participants 2 Years to Less Than 18 Years of Age With Moderately to Severely Active Ulcerative Colitis
Brief Title: A Study of Mirikizumab (LY3074828) in Pediatric Participants With Moderately to Severely or Active Ulcerative Colitis
Acronym: SHINE-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16634; I6T-MC-AMBA (Other: Eli Lilly and Company); 2022-502183-20-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-03-13; First posted 2023-03-24 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — mirikizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Mirikizumab Weight-Based Group 1 (Experimental): Experimental: Participants will receive mirikizumab weight-based dosing intravenously (IV) or subcutaneously (SC).
  Interventions: Drug: Mirikizumab IV; Drug: Mirikizumab SC
- Mirikizumab Weight-Based Group 2 (Experimental): Experimental: Participants will receive mirikizumab weight-based dosing IV or SC.
  Interventions: Drug: Mirikizumab IV; Drug: Mirikizumab SC
- Mirikizumab Weight-Based Group 3 (Experimental): Experimental: Mirikizumab Participants will receive mirikizumab weight-based dosing IV or SC.
  Interventions: Drug: Mirikizumab IV; Drug: Mirikizumab SC

INTERVENTIONS:
Drug: Mirikizumab IV — Administered IV
  Other Names: LY3074828
Drug: Mirikizumab SC — Administered SC
  Other Names: LY3074828

SUMMARY:
The main purpose of this study is to investigate efficacy, pharmacokinetics and safety of the drug in pediatric participants with moderately to severely active ulcerative colitis (UC).

DETAILED DESCRIPTION:
Participants who complete the study will have the option to enter the long-term extension Study I6T-MC-AMAZ (AMAZ).

ELIGIBILITY:
Inclusion Criteria:

* Males or females weighing ≥10 kg and ≥2 and <18 years old at the time of consent for screening.
* Have moderate to severe UC.
* Have failed corticosteroids, biologics, (for example, anti-tumor necrosis factor (TNF) antibodies or anti-integrin antibodies), immunomodulators (for example, azathioprine, thiopurines or methotrexate) or Janus Kinase (JAK)-Inhibitor treatment.
* Have UC at least 3 months in duration before baseline, which includes endoscopic evidence of UC corroborated by a histopathology report.

Exclusion Criteria:

* Have Crohn's disease, Inflammatory Bowel Disease Unclassified, ulcerative proctitis or primary sclerosing cholangitis.
* Have immune deficiency syndrome.
* Previous bowel resection or intestinal surgery.
* Evidence of toxic megacolon.
* History or current evidence of cancer of the gastrointestinal tract.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with modified Mayo score (MMS) Clinical Remission at Week 52 among the Week 12 Clinical Responders | Baseline to Week 52

SECONDARY OUTCOMES:
Percentage of Participants in MMS Clinical Remission | Week 12
Percentage of Participants in MMS Clinical Response | Week 12
Percentage of Participants with Endoscopic Remission | Week 12
Percentage of Participants with Endoscopic Improvement | Week 12
Percentage of Participants Achieving Pediatric Ulcerative Colitis Activity Index (PUCAI) Clinical Response | Week 12
Percentage of Participants Achieving PUCAI Clinical Remission | Week 12
Percentage of Participants Achieving Histologic Endoscopic Mucosal Improvement | Week 12
Percentage of Participants Achieving MMS Clinical Response | Week 52
Percentage of Participants Achieving MMS Clinical Remission | Week 52
Percentage of Participants Achieving PUCAI Clinical Response | Week 52
Percentage of Participants Achieving PUCAI Clinical Remission | Week 52
Percentage of Participants Achieving Endoscopic Remission | Week 52
Percentage of Participants Achieving Endoscopic Improvement | Week 52
Percentage of Participants Achieving MMS Clinical Remission without Surgery at Week 52 among Clinical Responders at Week 12 and without the Use of Corticosteroids | Baseline to Week 52
Percentage of Participants Achieving Histologic Endoscopic Mucosal Improvement | Week 52
Pharmacokinetics (PK): Area Under the Curve (AUC) of Mirikizumab | Baseline to Week 52
  PK: AUC of Mirikizumab
PK: Cmax of Mirikizumab | Baseline to Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (6):
  - University of California, San Francisco, San Francisco, California
  - Children's Center for Digestive Health Care, LLC, Atlanta, Georgia
  - Riley Childrens Hospital, Indianapolis, Indiana
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
- Belgium (2):
  - UZA, Edegem
  - UZ Leuven, Leuven
- The Hospital for Sick Children, Toronto, Canada
- Hôpital Necker - Enfants Malades, Paris, France
- Germany (3):
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz
  - LMU-Campus Innenstadt, München
  - Helios Klinikum Wuppertal, Wuppertal
- Israel (4):
  - Shaare Zedek, Jerusalem
  - Hadassah University Hospital, Ein Kerem, Jerusalem
  - Schneider Children's Medical Center, Petah Tikva
  - King Fahad Medical City, Rishon LeZiyyon
- Italy (2):
  - Azienda Ospedaliero Universitaria Ospedale Pediatrico Meyer, Florence
  - Azienda Ospedaliera Universitaria Policlinico Umberto I - Università di Roma La Sapienza, Roma
- Japan (6):
  - Juntendo University Hospital, Bunkyō City
  - Institute of Science Tokyo Hospital, Bunkyō City
  - Kokikai Tsujinaka Hospital Kashiwanoha, Kashiwa-shi
  - Saga University Hospital, Saga
  - National Center for Child Health and Development, Setagaya-ku
  - Yokohama City University Medical Center, Center of IBD, Yokohama
- Poland (5):
  - Gabinet Lekarski Bartosz Korczowski, Rzeszów
  - Twoja Przychodnia-Szczecińskie Centrum Medyczne, Szczecin
  - Medical Network Spółka z o. o., WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Instytut 'Pomnik - Centrum Zdrowia Dziecka, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- South Korea (3):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Severance Hospital, Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Sheffield Children's Hospital, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Mirikizumab (LY3074828) in Pediatric Participants With Moderately to Severely or Active Ulcerative Colitis (SHINE-2) — https://trials.lilly.com/en-US/trial/395116